CLINICAL TRIAL: NCT07087041
Title: Prediction of Recompensation and Stable Recompensation in Patients With Decompensated Cirrhosis Using Spleen Stiffness Combined With Non-Invasive Markers: A Prospective, Observational, Multicenter Study
Brief Title: A Study to Predict Recompensation in Patients With Decompensated Cirrhosis Using Spleen Stiffness and Simple Blood Tests
Acronym: LEAD-2
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hong You, Dr, Beijing Friendship Hospital
Other Study IDs: 2025-P2-244-01
Record Dates: First submitted 2025-07-04; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Decompensated Cirrhosis; Hepatitis B Virus (HBV) Infection; Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD); Alcohol-Related Liver Disease; Portal Hypertension; Recompensation
Keywords: Recompensation; Decompensated Cirrhosis; Spleen Stiffness
MeSH Terms: conditions — Hepatitis B; Infections; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recompensation group: ≥12 months since the last decompensated event
- Non-recompensation group: <12 months since the last decompensated event

SUMMARY:
The goal of this observational study is to learn if spleen stiffness and other non-invasive markers can help predict recompensation in people with decompensated cirrhosis who are receiving effective treatment for the cause of their liver disease. The main questions it aims to answer are:

* Can spleen stiffness and blood test results predict who will get better and stay better after cirrhosis becomes worse?
* What are the features of people who recover after decompensation?

Participants will:

* Be people with decompensated cirrhosis who are already getting effective treatment (such as antiviral therapy or alcohol abstinence)
* Be followed over time to check if they remain stable or have more liver problems
* Have non-invasive tests done, including spleen stiffness measurement and blood tests

Researchers will track how many participants recover and stay recovered over time, and use that information to build a tool to help predict outcomes in others with cirrhosis.

DETAILED DESCRIPTION:
This is a prospective, observational, multicenter study designed to follow adults with decompensated cirrhosis who are receiving effective treatment for the underlying cause of their liver disease, such as antiviral therapy, alcohol abstinence, or metabolic management. The study is aiming to understand how these patients recover after treatment; Identify how often they achieve recompensation and stable recommendation; Develop a non-invasive model using spleen stiffness and other markers to predict who is more likely to improve.

Participants will be grouped based on whether they have had decompensation within the past 12 months. Researchers will regularly collect clinical data, spleen stiffness measurements, and lab tests, to develop and validate a model that predicts recompensation and stable recompensation. The study will also assess the cumulative incidence of clinical events (e.g., further decompensation, hepatocellular carcinoma, liver transplantation, and death) over a two-year follow-up period. Predictive accuracy, model calibration, and discrimination will be evaluated using standard statistical methods, including competing risk models and AUROC analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 75 years (inclusive)
* Clinically diagnosed decompensated cirrhosis
* First decompensated event occurred within 12 months of screening, or no decompensated events in the past 12 months despite a history of decompensation
* Received effective etiological treatment per guidelines:

  * For HBV: Sustained antiviral suppression
  * For alcohol-related liver disease: Sustained abstinence for ≥2 months
  * For MAFLD-related cirrhosis: Improved liver function after lifestyle/ metabolic intervention

Exclusion Criteria:

* Missing data on first decompensated event
* Prior orthotopic liver transplantation or TIPS
* Prior splenectomy, splenic embolization, or other shunt surgery
* History or current diagnosis of hepatocellular carcinoma
* Acute variceal bleeding within the last 4 weeks or unstable condition
* Uncontrolled moderate-to-severe ascites
* Cholestatic cirrhosis; untreated chronic liver diseases; non-cirrhotic portal hypertension; vascular liver diseases (e.g., Budd-Chiari syndrome)
* Acute or chronic portal vein thrombosis
* Severe comorbidities of heart, lung, kidney, brain, hematologic, or psychiatric systems
* Other systemic malignancies (except cured cases)
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 75 years with decompensated cirrhosis who are receiving and maintaining effective treatment for the underlying cause of liver disease. The first decompensation event must be clinically significant ascites and/or variceal bleeding. Participants must have either experienced their first decompensation within the past 12 months or remained free from new decompensation events during the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 735 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of non-invasive models based on spleen stiffness in predicting Recompensation | 2 years
  The primary outcome of this study is the accuracy of a non-invasive prediction model based on spleen stiffness and routine laboratory markers in identifying recompensation and stable recompensation in individuals with decompensated cirrhosis.

SECONDARY OUTCOMES:
Discrimination, calibration, and stability of the prediction model | 2 years
  This outcome assesses the performance of the prediction model developed to identify recompensation and stable recompensation in people with decompensated cirrhosis.
Predictive accuracy of spleen stiffness in identifying recompensation and stable recompensation | 2 years
  This outcome evaluates the predictive accuracy of spleen stiffness in identifying recompensation and stable recompensation among participants with decompensated cirrhosis.
Predictive accuracy of liver stiffness in identifying recompensation and stable recompensation | 2 years
  This outcome evaluates the predictive accuracy of liver stiffness in identifying recompensation and stable recompensation among participants with decompensated cirrhosis.
Predictive accuracy of platelets in identifying recompensation and stable recompensation | 2 years
  This outcome evaluates the predictive accuracy of platelet count in identifying recompensation and stable recompensation among participants with decompensated cirrhosis.
Cumulative incidence of recompensation by etiology | 2 years
  This outcome measures the 2-year cumulative incidence of recompensation among participants with decompensated cirrhosis, stratified by the underlying cause of liver disease (etiology). Recompensation is defined as the effective control or removal of the primary cause of liver disease, resolution of ascites and hepatic encephalopathy with no episodes of variceal bleeding for at least 12 months, and improvement in liver function indicated by a Child-Pugh classification of Class A and/or a MELD score below 10.
Cumulative incidence of stable recompensation by etiology | 2 years
  This outcome measures the 2-year cumulative incidence of stable recompensation in participants with decompensated cirrhosis, stratified by liver disease etiology. Stable recompensation is defined as achieving recompensation and maintaining that status without further decompensated events for at least one additional year.
Cumulative incidence of further decompensation by etiology | 2 years
  This outcome evaluates the 2-year cumulative incidence of further decompensation among participants with decompensated cirrhosis, stratified by the underlying etiology of liver disease. Further decompensation is defined as the occurrence of new or worsening clinical events such as ascites, hepatic encephalopathy, or variceal bleeding after initial enrollment.
Cumulative incidence of liver-related composite endpoints by etiology | 2 years
  This outcome assesses the 2-year cumulative incidence of liver-related composite endpoints among participants with decompensated cirrhosis, stratified by liver disease etiology.Liver-related composite endpoints include the first occurrence of any of the following events: Further hepatic decompensation (e.g., ascites, variceal bleeding, hepatic encephalopathy); Hepatocellular carcinoma (HCC); Liver transplantation; Liver-related death.

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, Prof., Principal Investigator — Beijing Friendship Hospital
Locations (28):
- China (28):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Foshan Traditional Chinese Medicine Hospital, Foshan, Guangdong
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Panyu Central Hospital, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Zhuhai, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Taihe Hospital, Shiyan, Shiyan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Nanjing Second Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Huadong Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Jincheng People's Hospital, Jincheng, Shanxi
  - Jinzhong People's Hospital, Jinzhong, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data to be shared include de-identified demographic information, clinical characteristics, laboratory test results (including spleen stiffness, liver stiffness, platelet counts, and other routine blood tests), treatment details, and clinical outcomes related to recompensation and stable recompensation.
Supporting Information: Study Protocol, CSR
Time Frame: Individual participant data (IPD) and supporting documentation will be available beginning 6 months after publication of the primary study results.
Access Criteria: Qualified researchers affiliated with academic or medical institutions will be able to request access to the de-identified individual participant data (IPD) and supporting documents (such as study protocol and statistical analysis plan).
  All requests will be reviewed and approved by the study steering committee.
URL: https://www.clinicaltrials.gov/